CLINICAL TRIAL: NCT05126394
Title: A Comparative Study Between Ultrasound-guided Serratus Anterior Plane Block and Conventional IV Analgesics in Postoperative Pain Management in Modified Radical Mastectomy
Brief Title: U/S Guided SAPB Versus Conventional IV Analgesics in Postoperative Pain Management in MRM
Acronym: SAPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MD 209a / 2021
Record Dates: First submitted 2021-10-26; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2020-03

CONDITIONS: Injection Site Haematoma; Local Anesthetic Toxicity
Keywords: "SAPB"; "MRM"; "pain management"
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled clinical trial.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A ( SAPB) group (Experimental): this group of patients receives serratus anterior plane block, just after induction of anesthesia.
  Interventions: Procedure: ultrasound guided serratus anterior plane block
- Group B: control group (No Intervention): this group of patients does not receive any blockade, they receive conventional IV analgesics.

INTERVENTIONS:
Procedure: ultrasound guided serratus anterior plane block — the patients receive local anesthetic (20 ml of Bupivacaine 0.25 %), injected superficial to the serratus muscle under ultrasound guidance.
  Arms: Group A ( SAPB) group

SUMMARY:
The aim of this study is to compare the effect of ultra-sound guided serratus anterior plane block versus conventional IV analgesics in postoperative pain management in modified radical mastectomy (MRM)

DETAILED DESCRIPTION:
All patients undergoing modified radical mastectomy were assigned to one of the following two groups:Group A: Serratus anterior plane block group (SAPB group): this group consists of 20 patients who received ultra sound guided serratus anterior plane block just after induction of anesthesia and Group B: IV analgesics group (control group): this group consists of 20 patients who did not receive any type of block.Further evaluations were carried out by a different investigator who was unaware of the patients' grouping. The degree of post-operative pain was assessed at: just upon arrival to the PACU, 2, 4, 8, 12 and 24 hours using the VAS score and the haemodynamic data and respiratory rate were measured during the first 24 hours after the end of the surgery. Postoperative analgesia regimen was standard in both groups; patients from each groups received 1 gm of Paracetamol Q 8 hours.

Patients reporting VAS ( visual analogue score) score greater than 40, mean arterial blood pressure, heart rate or respiratory rate >20% from the baseline, were given Pethidine (50 mg IV) as rescue analgesic. While, those reporting VAS score less than 40 with mean arterial blood pressure, heart rate or respiratory rate >20% from the baseline but still complaining; Ketoralac (30 mg IV) was given with a maximum dose of 120 mg/ day.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 20-60 years old.
* Preoperative physical status: ASA (American Society of Anesthesiology) I & II.
* Body mass index (BMI) < 35 Kg/ m2.
* Candidate for unilateral modified radical mastectomy.
* Informed consent to participate in the study.

Exclusion Criteria:

* - Females aged < 20 years old or > 60 years old.
* Preoperative physical status: ASA III & IV.
* Morbid obese patients with BMI > 35 Kg/ m2.
* Refusal to participate in the study.
* Addiction to narcotics or psycho-active drugs.
* Psychological disorders.
* Contra-indications to regional anesthesia (coagulopathy, injection site infection or allergy to any of the study drugs)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
the time of first rescue analgesic | it is measured for 24 hours after the end of surgery.
  the time taken by the patient to receive first dose of rescue analgesia, guided by the patients VAS score ( if the patients VAS score is 4 or more, the patient receives 50 mg of Pethidine).
total dose of rescue analgesics | it is measured for 24 hours after the end of surgery.
  the total dose of Pethidine needed by each patient measured in mg.

SECONDARY OUTCOMES:
patients satisfaction | 24 hours after the end of surgery.
  patients satisfaction is measured on a scale from 0 to 10, where 0 means not satisfied at all and 10 means the ultimate satisfaction.
incidence of nausea and vomiting | 24 hours after the end of surgery.
  patients are assessed for incidence of postoperative nausea and vomiting.
incidence of any block related complications. | 24 hours after the end of surgery.
  incidence of any serratus anterior plane block complications (e.g. injection site hematoma, signs and/or symptoms of local anesthetic toxicity ) is detected.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Gomaa Salama, Medical Doctorate, Study Director — Anesthesia department, Ain Shams University, Cairo, Egypt.; Hanan Mahmoud Farag, Medical Doctorate, Study Director — Anesthesia department, Ain Shams University, Cairo, Egypt.
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt